CLINICAL TRIAL: NCT06509178
Title: The Effect of Two dıfferent Teaching Approaches in Nursing Skills Training on Objective Performance, Self-regulated Learning and Satisfaction
Brief Title: The Effect of Two Different Teaching Approaches in Nursing Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, özlem doğu, Associate Professor Doctor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Peyton and Halsted Method
Record Dates: First submitted 2024-07-10; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Urinary Retention
Keywords: Urinary Catheterization; Peyton Model; Halsted Model; Laboratory Applications
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Two randomized control group. One applied Halsted , other applied Peyton 4-step model on nursing students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peyton group (Experimental): The experimental group students attended the course in accordance with the routine procedures but in the laboratory practice, sterile urinary catheter application was taught to the students according to Peyton's 4-step approach.
  In the first stage of the method, students were only asked to watch the researcher demonstrate the application.
  In the second step, the sterile urinary catheterization process was demonstrated a second time by the researcher, with each step explained in detail.
  In the third step, the students were asked to give guidance and repeat the steps while the researcher applied the application for the third time.
  In the fourth step, each student was asked to perform the application individually without any help.
  Interventions: Other: Peyton group
- Halsed group (Other): The control group students attended the course in accordance with the routine procedures, students were taught how to apply sterile urinary catheter using the Halsted method (see one and do it), which is traditionally used in laboratory practice.
  Interventions: Other: Halsed group

INTERVENTIONS:
Other: Peyton group — The same procedures were applied to the students in the experimental group as the students in the control group, except for laboratory applications. Students were asked to watch the video contents after the theoretical course, and in the laboratory practice, sterile urinary catheter application was taught to the students according to Peyton's 4-step approach. Before the skill demonstration, students were given information about the research. Students were given 15-20 minutes to fill out the voluntary consent form and the urinary catheterization success pre-test. Students were taught the sterile urinary catheter procedure in accordance with Peyton's 4-step approach.The research was conducted on the days and hours of the students' laboratory days. The data collection phase of the research took 3 weeks in total.
  Arms: Peyton group
Other: Halsed group — After the control group students attended the course in accordance with the routine procedures, the students were asked to watch videos of the online urinary catheter application course and the students were taught how to apply sterile urinary catheter using the Halsted method (see one and do it), which is traditionally used in laboratory practice. Students were informed about the research and voluntary consent forms were obtained. Students were given 15-20 minutes to complete the urinary catheterization success pre-test. During the demonstration, the students' questions were answered, the researcher went over the points that the student did not understand, corrected any incorrect behavior, and gave feedback. Afterwards, each student was asked to demonstrate the skill steps individually.The research was conducted on the days and hours of the students' laboratory days. The data collection phase of the research took 3 weeks in total.
  Arms: Halsed group

SUMMARY:
The purpose of this study is effectiveness of Peyton 4-step teaching method and Halsted method on nursing students. The research was conducted as a randomized controlled experimental study with first-year nursing students on urinary catheter within the scope of the Nursing Fundamentals course of Sakarya University Health Sciences Institute. The result of Personal Information Form, Self-Directed Learning Scale in Clinical Nursing Practice, Stress and Satisfaction Vas Scale, Urinary Catheterization Success Pre and Post-Test and Urinary Catheter Application Skill Checklist were comperisoned.

DETAILED DESCRIPTION:
Nursing is a discipline where teaching clinical skills is extremely important. In addition to the traditional methods used in laboratory practices in nursing, the use of innovative methods contributes to learning. This research was conducted experimentally to evaluate the effectiveness of the Peyton and Halsted teaching method in nursing student's urinary catheterization skill learning.

The research was conducted as a randomized controlled experimental study with first-year nursing students within the scope of the Nursing Fundamentals course of Sakarya University Health Sciences Institute in the spring semester of the 2022-2023 academic year. The sample of the study consisted of 217 randomly selected students, 108 students in the experimental group and 109 students in the control group. In the research, Peyton's 4-step teaching method was applied to the experimental group during urinary catheterization laboratory applications. For the control group, the traditional Halsted method was used. Data were collected with the Personal Information Form, Self-Directed Learning Scale in Clinical Nursing Practice, Stress and Satisfaction Vas Scale, Urinary Catheterization Success Pre- and Post-Test, and Urinary Catheter Application Skill Checklist. The knowledge and skills learning levels of the experimental and control group students were compared. Descriptive statistics, Pearson chi-square, Mann-Whitney U and Kruskal Wallis tests were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* First year student at the Faculty of Nursing,
* Enrolling in the "Fundamentals of Nursing" course for the first time,
* Have watched the video recordings of the online application of Sakarya University Faculty of Health Sciences SAÜSEM (Sakarya University Continuing Education Application and Research Center),
* Students who agreed to participate in the research

Exclusion Criteria:

* Graduate of health vocational high school,
* Settled through the foreign student exam (YÖS),
* After graduating from the fields that provide associate degree education related to health, they were placed in the nursing department with the vertical transfer exam (DGS),
* Students who take the "Fundamentals of Nursing" course as a repeat

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Urinary catheter application skill checklist | 3 weeks
  It was used to measure to what extent the student learned the skill after the skill laboratory training. It is a list consisting of 40 items containing skill check steps for urinary catheterization and used by the researcher during the evaluation phase of the student with the Objective Structured Clinical Examination (OSCE) method. While preparing the list, a literature review was conducted, existing laboratory application books were used, and expert opinions were taken. Content validity indexes were calculated using the Davis Technique.

SECONDARY OUTCOMES:
Urinary Catheterization Achievement Knowledge Test | 3 weeks
  To determine the students' knowledge level on the subject before the laboratory application, their knowledge level on the subject to be taught was measured by testing before and after the application. The test was re-evaluated before and after application. In the preparation of the success pre- and post-tests, questions were prepared by reviewing the literature on the subject and taking expert opinions. The application of urinary catheterization was created from 20 questions involving laboratory skills and expert opinions were taken
Self-Regulated Learning Scale for Clinical Nursing Practice | 3 weeks
  he scale used in the study was developed by Satoko Iyama and Hitomi Maeda (Iyama & Maeda, 2018) in 2017. The Turkish validity and reliability of the scale was conducted by Şenol (2018). It has been reported that the scale is valid and reliable for nursing students (Şenol, 2018). The scale consists of 16 items. The scale has two sub-dimensions: "Motivation" and "Learning Strategies". The lowest score that can be obtained from this Scale is 16 and the highest score is 80. As the score obtained from the scale increases, the student's use of the self-regulated learning approach increases.
Satisfaction and stress level | 3 weeks
  Measured using the Visual Analog Scale (VAS) and numbering method from one to ten. In determining the level, "0" indicated dissatisfaction and no stress, while "10" indicated very satisfied and high stress.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Doğu, Study Director — Sakarya University Faculty of Health Sciences
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No